CLINICAL TRIAL: NCT04551703
Title: The Effect of Intranasal Irrigation With Adrenaline Solution on Intraoperative Visualization and Bleeding During Functional Endoscopic Sinus Surgery
Brief Title: Adrenaline Solution Irrigation and Bleeding During Sinus Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 221
Record Dates: First submitted 2020-08-23; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
Keywords: Sinusitis; Nasal Polyp; Endoscopic Sinus Surgery; Adrenaline
MeSH Terms: conditions — Disease; Sinusitis; Nasal Polyps

STUDY DESIGN:
Intervention Model Description: Patients will randomize into two groups based on computer generating numbers. Group 1 will have the usual method of irrigation with normal saline during surgery whereas group 2 have irrigation with 1:100 000 adrenaline in normal saline. The solution will be prepared by the senior resident through adding one ampule of 0.1 percent adrenaline in one liter bag of normal saline, which made the adrenaline concentration in the solution 1:100 000. The investigators who collected the data will be blinded to the content of both preparations. Irrigation with either solution will be used during the procedure through a 20 mL syringe attached to an olive tip long curved suction.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adrenaline saline irrigation (Experimental): Adrenaline saline irrigation will be prepared by adding one ampule of 0.1 percent adrenaline in one liter bag of normal saline, which made the adrenaline concentration in the solution 1:100 000
  Interventions: Drug: Adrenaline saline irrigation
- Normal saline irrigation (No Intervention): Normal saline bag will be used for irrigation during the procedure

INTERVENTIONS:
Drug: Adrenaline saline irrigation — The surgical field is flushed with 20 cc of Adrenaline saline irrigation. This is in contrast to the standard of care, normal saline irrigation.
  Other Names: Epinephrine saline irrigation
  Arms: Adrenaline saline irrigation

SUMMARY:
Intranasal irrigation with normal saline is routinely used in sinus surgery to clean the tip of the nasal endoscope and clear the surgical field from blood. The purpose of this study is to evaluate the difference in the surgical visualization, surgeon satisfaction and total blood loss when intraoperative irrigation was performed with a solution of normal saline with adrenaline as compared to irrigation with normal saline alone in FESS.

DETAILED DESCRIPTION:
Functional Endoscopic Sinus Surgery (FESS) is a common, effective and minimally invasive surgical procedure indicated mainly to treat medically resistant chronic rhinosinusitis with or without nasal polyposis.

The surgery is often performed under general anesthesia and proceeds in anatomically based surgical landmarks steps to facilitate drainage and ventilation of the paranasal sinuses. As any other endoscopic and laparoscopic procedures the operation requires dry surgical field to ensure accurate identification and visualization of structures and smooth surgical dissection progression. Intranasal bleeding during FESS will increase time of surgery and perioperative complications. Also it could affect healing process, increase adhesion formation and lengthening recovery period .

Different methods and maneuvers have been described in the literature to reduce intra-operative bleeding during sinus surgery. These include: elevation of the patient's head, the use of bipolar cautery and powered instruments; premedication with beta blockers; a controlled hypotensive anesthesia technique; total intravenous anesthesia, topical hemostatic biomaterials and local application of vasoconstrictors.

Adrenaline is one of the most commonly used topical vasoconstrective agent. Because systemic absorption of infiltrated adrenaline can give rise to a sudden increase in blood levels of catecholamine compared to topical instillation and thus various life-threatening complications, such as : cardiac arrhythmia, cardiac arrest, cardiomyopathy, pulmonary edema, and central retinal artery occlusion; many surgeons prefer to use instillation of adrenaline over infiltration in FESS

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologist (ASA) classification <2
* Patients with chronic with or without nasal polyposis refractory to medical treatment

Exclusion Criteria:

* Patients with a history of of bleeding diathesis
* Patients with severe ischemic heart disease , pulmonary and renal disease
* Patients with tumours or vascular anomalies
* Patients with cystic fibrosis, allergic fungal sinusitis and granulomatous disorders
* Patients who are unable to speak, read and write English

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
The Boezaart intraoperative surgical field scale | 2 hours
  The Boezaart intra-operative surgical field scale will be used to grade the level of bleeding during surgery. This 0 to 5-point scale will be used to outline the amount of suction required to rid the area of blood disrupting vision. A score of 0 is given for an area with no bleeding, 1 for slight bleeding with no suction required, 2 for slight bleeding requiring suction, 3 for moderate bleeding which improves for several seconds once suction has occurred, 4 for moderate bleeding which restarts directly after suctioning and 5 for severe bleeding which occurs faster then can be removed

SECONDARY OUTCOMES:
Volume of total blood loss | The volume of blood loss will be measured every 30 minutes from the start of surgery for the duration of 2 hours
  Total blood loss will be calculated and measured over the duration of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Mohannad A Al-Qudah, MD,FACS, Study Chair — Jordan University of Science & Technology & King Abdullah University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Higgins TS, Hwang PH, Kingdom TT, Orlandi RR, Stammberger H, Han JK. Systematic review of topical vasoconstrictors in endoscopic sinus surgery. Laryngoscope. 2011 Feb;121(2):422-32. doi: 10.1002/lary.21286. Epub 2011 Jan 13. PMID 21271600
- [Result] Saif AM, Farboud A, Delfosse E, Pope L, Adke M. Assessing the safety and efficacy of drugs used in preparing the nose for diagnostic and therapeutic procedures: a systematic review. Clin Otolaryngol. 2016 Oct;41(5):546-63. doi: 10.1111/coa.12563. Epub 2016 Feb 11. PMID 26452438
- [Result] Yim MT, Ahmed OG, Takashima M. Evaluating real-time effects of topical 1:1000 epinephrine in endoscopic sinus and skull-base surgery on hemodynamic parameters through intraoperative arterial line monitoring. Int Forum Allergy Rhinol. 2017 Nov;7(11):1065-1069. doi: 10.1002/alr.22012. Epub 2017 Sep 18. PMID 28922579
- [Result] Khosla AJ, Pernas FG, Maeso PA. Meta-analysis and literature review of techniques to achieve hemostasis in endoscopic sinus surgery. Int Forum Allergy Rhinol. 2013 Jun;3(6):482-7. doi: 10.1002/alr.21126. Epub 2012 Dec 16. PMID 23255493
- [Result] Gan EC, Alsaleh S, Manji J, Habib AR, Amanian A, Javer AR. Hemostatic effect of hot saline irrigation during functional endoscopic sinus surgery: a randomized controlled trial. Int Forum Allergy Rhinol. 2014 Nov;4(11):877-84. doi: 10.1002/alr.21376. Epub 2014 Aug 18. PMID 25137523